CLINICAL TRIAL: NCT04601051
Title: Phase 1 Two-Part (Open-label, Single Ascending Dose (Part 1) and Open-label, Single Dose Expansion (Part 2)) Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NTLA-2001 in Patients With Hereditary Transthyretin Amyloidosis With Polyneuropathy (ATTRv-PN) and Patients With Transthyretin Amyloidosis-Related Cardiomyopathy (ATTR-CM)
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NTLA-2001 in Patients With Hereditary Transthyretin Amyloidosis With Polyneuropathy (ATTRv-PN) and Patients With Transthyretin Amyloidosis-Related Cardiomyopathy (ATTR-CM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ITL-2001-CL-001; 2020-002034-32 (EudraCT Number)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy; Transthyretin-Related (ATTR) Familial Amyloid Cardiomyopathy; Wild-Type Transthyretin Cardiac Amyloidosis
Keywords: NTLA-2001; Pharmacokinetics; Pharmacodynamics; Neurologic Function; Clustered Regularly Interspaced Short Palindromic Repeats; CRISPR; Polyneuropathy; ATTR; Transthyretin; TTR; Amyloidosis; Familial Amyloid Polyneuropathy; FAP; Cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Polyneuropathies; Amyloidosis; Cardiomyopathies | interventions — NTLA-2001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Polyneuropathy Part 1: NTLA-2001 (Experimental): Participants, assigned to one of 4 dose-escalation cohorts, will receive a single dose of NTLA-2001.
  Interventions: Biological: NTLA-2001
- Polyneuropathy Part 2: NTLA-2001 (Experimental): Participants, assigned to the dose-expansion cohort, will receive a single dose of NTLA-2001.
  Interventions: Biological: NTLA-2001
- Cardiomyopathy Part 1 (UK only): NTLA-2001 (Experimental): Participants, assigned to one of 2 dose-escalation cohorts, will receive a single dose of NTLA-2001.
  Interventions: Biological: NTLA-2001
- Cardiomyopathy Part 2 (UK only): NTLA-2001 (Experimental): Participants, assigned to the dose-expansion cohort, will receive a single dose of NTLA-2001.
  Interventions: Biological: NTLA-2001
- Polyneuropathy Follow-on Dosing (PN Part 1 Dose Level 1 Subjects only): NTLA-2001 (Experimental): Participants assigned to the follow-on dosing cohort will receive a subsequent dose of NTLA-2001.
  Interventions: Biological: NTLA-2001

INTERVENTIONS:
Biological: NTLA-2001 — A clustered regularly interspaced short palindromic repeats (CRISPR)/Cas9 gene editing system delivered by lipid nanoparticles (LNPs) for intravenous (IV) administration

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of NTLA-2001 in participants with hereditary transthyretin amyloidosis with polyneuropathy (ATTRv-PN) and participants with hereditary transthyretin amyloidosis with cardiomyopathy (ATTRv-CM) or wild type cardiomyopathy (ATTRwt-CM)

DETAILED DESCRIPTION:
For ATTRv-PN participants, Part 1 consists of an open-label, single-ascending dose study, which identifies the dose for evaluation in the cohort expansion of Part 2. Part 2 will follow as an open-label, dose expansion study to further characterize the activity of NTLA-2001, provide an initial assessment of the effect of NTLA-2001 on clinical measures of neuropathy and neurological function, and obtain additional safety data.

For ATTR-CM participants, Part 1 consists of an open-label, single-ascending dose study, which identifies the dose for evaluation in the cohort expansion of Part 2. Part 2 will follow as an open-label, dose expansion study to further characterize the activity of NTLA-2001, provide an initial assessment of the effect of NTLA-2001 on cardiac measures, and obtain additional safety data.

All participants who are dosed with NTLA-2001 will be offered to participate in a long-term safety monitoring follow-up study via a separate protocol.

ELIGIBILITY:
Polyneuropathy Inclusion Criteria:

* Male and/or female participants 18 to 80 years of age inclusive, at the time of signing the informed consent
* Diagnosis of polyneuropathy (PN) due to transthyretin (TTR) amyloidosis (ATTR)
* Must have a body weight of at least 45 kilograms (kg) at Screening visit
* Lack of access to approved treatments for ATTR and/or progression of hereditary transthyretin amyloidosis with polyneuropathy (ATTRv-PN) despite use of approved treatment for ATTRv-PN

Polyneuropathy Exclusion Criteria:

* Amyloidosis attributable to non-TTR protein, e.g., amyloid light-chain (AL) amyloidosis
* Known leptomeningeal transthyretin amyloidosis
* Use of any of the following TTR-directed therapy for ATTR within certain timeframe:

  1. Patisiran
  2. Inotersen
  3. Vutrisiran
  4. Tafamidis
  5. Diflunisal
  6. Doxycycline and/or tauroursodeoxycholic acid
  7. Any other investigational agent for the treatment of ATTRv-PN:
* Other protocol defined Inclusion/Exclusion criteria may apply

Cardiomyopathy Inclusion Criteria (UK only):

* Male and/or female participants 18 to 90 years of age inclusive, at the time of signing the informed consent
* Diagnosis of transthyretin (ATTR) amyloidosis with cardiomyopathy, classified as hereditary ATTR amyloidosis with cardiomyopathy (ATTRv-CM) or wild type cardiomyopathy (ATTRwt-CM).
* Must have a body weight of at least 45 kilograms (kg) at Screening visit
* New York Heart Association (NYHA) Class I-III heart failure
* At least 1 prior hospitalization for heart failure and/or clinical evidence of heart failure.
* Able to complete ≥150 meters on the 6-minute walk test (6-MWT) during the Screening period.

Cardiomyopathy Exclusion Criteria (UK only):

* Amyloidosis attributable to non-TTR protein, e.g., amyloid light-chain (AL) amyloidosis
* Known leptomeningeal transthyretin amyloidosis
* Use of any of the following TTR-directed therapy for ATTR within certain timeframes:

  1. Patisiran
  2. Inotersen
  3. Vutrisiran
  4. Tafamidis
  5. Diflunisal
  6. Doxycycline and/or tauroursodeoxycholic acid
  7. Investigational TTR stabilizer (e.g., AG-10)
* Participants with heart failure that in the opinion of the investigator is caused by ischemic heart disease, hypertension, or uncorrected valvular disease and not primarily due to transthyretin amyloid cardiomyopathy.
* Participants with a history of sustained ventricular tachycardia or aborted ventricular fibrillation or with a history of atrioventricular (AV) nodal or sinoatrial (SA) nodal dysfunction for which a pacemaker is indicated but will not be placed. Pacemaker or defibrillator placement, initiation of or change in anti-arrhythmic medication within 28 days prior to study drug administration.
* Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events | up to Day 730
Number of Participants with Clinically Significant Clinical Laboratory Test Findings | up to Day 730
Number of Participants with Clinically Significant Safety Measurements | up to Day 730
Percent Change from Baseline in Serum TTR (enzyme-linked immunosorbent assay [ELISA]) | up to Day 730
Percent Change from Baseline in Serum Prealbumin | up to Day 730
Mean Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Measurable Concentration (AUClast) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Mean Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUCinf) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Mean Maximum Concentration (Cmax) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Mean Time of the Maximum Concentration (Tmax) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Mean Terminal Half-Life (t½) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Mean Apparent Clearance (CL) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Mean Volume of Distribution (Vd) for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | up to Day 730
Change from Baseline in Anti-Drug Antibody to NTLA-2001 and Anti-Cas9 Protein Antibody to Transgene Product Levels | up to Day 730

SECONDARY OUTCOMES:
Polyneuropathy only: Change from Baseline in Familial Amyloid Polyneuropathy (FAP) Stage. | up to Day 730
Polyneuropathy only: Change from Baseline in Polyneuropathy Disability (PND) Score | up to Day 730
Polyneuropathy only: Change from Baseline in Modified Body Mass Index (mBMI) | up to Day 730
Polyneuropathy only: Change from Screening in Neuropathy Impairment Score (NIS) | up to Day 730
Polyneuropathy only: Change from Baseline in Modified Neuropathy Impairment Score +7 (mNIS+7) | up to Day 730
Polyneuropathy only: Change from Screening in 10-Meter Walk Test (10-MWT) | up to Day 730
Polyneuropathy only: Change from Baseline in Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) | up to Day 730
Polyneuropathy only: Change from Baseline in EuroQOL (EQ)-5D-5L | up to Day 730
Cardiomyopathy only: Change from Baseline in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | up to Day 730
Cardiomyopathy only: Change from Baseline in hs Troponin T | up to Day 730
Cardiomyopathy only: Change from Baseline in Magnetic resonance imaging (MRI) | up to Day 730
Cardiomyopathy only: Change from Baseline in Echocardiogram | up to Day 730
Cardiomyopathy only: Change from Baseline in Cardio-pulmonary exercise test | up to Day 730
Cardiomyopathy only: Change from Baseline in 6-Minute Walk Test (6-MWT) | up to Day 730
Cardiomyopathy only: Change from Baseline in New York Heart Association (NYHA) Classification | up to Day 730
Cardiomyopathy only: Change from Baseline in Patient-reported outcomes (KCCQ) | up to Day 730

CONTACTS AND LOCATIONS:
Locations (4):
- Clinical Trial Site, Paris, France
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Umeå, Sweden
- Clinical Trial Site, London, United Kingdom

REFERENCES:
- [Derived] Gillmore JD, Gane E, Taubel J, Pilebro B, Echaniz-Laguna A, Kao J, Litchy W, Shahda S, Haagensen A, Walsh L, Smith D, Kachadourian J, Ward JH, Lebwohl D, Zhu P, Xu Y, Leung A, Sonderfan A, Gutstein DE, Manvelian G, Adams D. Nexiguran Ziclumeran Gene Editing in Hereditary ATTR with Polyneuropathy. N Engl J Med. 2025 Oct 9;393(14):1375-1386. doi: 10.1056/NEJMoa2510209. Epub 2025 Sep 25. PMID 41002250
- [Derived] Fontana M, Solomon SD, Kachadourian J, Walsh L, Rocha R, Lebwohl D, Smith D, Taubel J, Gane EJ, Pilebro B, Adams D, Razvi Y, Olbertz J, Haagensen A, Zhu P, Xu Y, Leung A, Sonderfan A, Gutstein DE, Gillmore JD. CRISPR-Cas9 Gene Editing with Nexiguran Ziclumeran for ATTR Cardiomyopathy. N Engl J Med. 2024 Dec 12;391(23):2231-2241. doi: 10.1056/NEJMoa2412309. Epub 2024 Nov 16. PMID 39555828
- [Derived] Gillmore JD, Gane E, Taubel J, Kao J, Fontana M, Maitland ML, Seitzer J, O'Connell D, Walsh KR, Wood K, Phillips J, Xu Y, Amaral A, Boyd AP, Cehelsky JE, McKee MD, Schiermeier A, Harari O, Murphy A, Kyratsous CA, Zambrowicz B, Soltys R, Gutstein DE, Leonard J, Sepp-Lorenzino L, Lebwohl D. CRISPR-Cas9 In Vivo Gene Editing for Transthyretin Amyloidosis. N Engl J Med. 2021 Aug 5;385(6):493-502. doi: 10.1056/NEJMoa2107454. Epub 2021 Jun 26. PMID 34215024
- [Derived] Stephenson AA, Flanigan KM. Gene editing and modulation for Duchenne muscular dystrophy. Prog Mol Biol Transl Sci. 2021;182:225-255. doi: 10.1016/bs.pmbts.2021.01.029. Epub 2021 Mar 3. PMID 34175043